CLINICAL TRIAL: NCT02828982
Title: Determining the Potential Benefit of Powered Prostheses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Deanna H Gates (Other)
Responsible Party: Sponsor-Investigator, Deanna H Gates, Assistant Professor, University of Michigan
Organization: University of Michigan (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: HUM00080734
Record Dates: First submitted 2016-06-29; First posted 2016-07-12 (Estimated); Results first posted 2020-11-13 (Actual); Last update posted 2022-01-18 (Actual); Status verified 2022-01

CONDITIONS: Unilateral Traumatic Amputation; Amputation, Traumatic
Keywords: powered ankle prosthesis; activity monitoring; muscle fatigue; below knee amputation
MeSH Terms: conditions — Amputation, Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Powered Ankle Prosthesis (Experimental): In this condition, the participant is fitted with a powered prosthetic ankle by a certified prosthetist. The ankle is the BiOM which is manufactured by Bionx (which used to be named iWalk). This device was given 510(K) Exempt status by the FDA under (regulation number: 890.3500). Participants will wear the device for 2 weeks.
  Interventions: Device: Powered ankle prosthesis
- Dynamic Response Foot (Sham Comparator): In this arm, participants will wear their clinically prescribed dynamic response foot. This period is 2 weeks long.
  Interventions: Device: Dynamic Response Foot

INTERVENTIONS:
Device: Powered ankle prosthesis — This device is a commercially available powered ankle prosthesis, (BioM, Bionx, Bedford, MA) which was given FDA device exempt status.
  Arms: Powered Ankle Prosthesis
Device: Dynamic Response Foot — This condition is a sham condition as the participant will wear the prosthesis they were clinically prescribed and usually wear.
  Arms: Dynamic Response Foot

SUMMARY:
The goal of this research is to determine the effectiveness of a powered prosthesis compared to an unpowered prosthesis during short bouts of walking, extended periods of walking (to fatigue), and performance in the community.

DETAILED DESCRIPTION:
Many individuals are living in the United States with limb loss. With the use of a prosthetic device many individuals can stay active, but most do not achieve a medically desired physical activity level. This creates a risk for cardiovascular disease. It is thought that individuals with amputation walk less because it is more difficult to get around, and recent advances in robotic prosthetic technology may make such activities easier. However, these prostheses have not yet been evaluated to determine their effectiveness during extended periods of walking. Despite the goals in design of new devices it is unclear whether individuals using them are able to incorporate them into making daily activities easier. Therefore, the goal of this research is to determine the effectiveness of a powered prosthesis compared to an unpowered prosthesis during long periods of walking.

ELIGIBILITY:
Inclusion Criteria:

* Adult (over 21 years old), Has unilateral transtibial amputation, has used prosthesis for at least 6 months, is currently using an unpowered prosthesis, can walk unassisted for at least 10 minutes

Exclusion Criteria:

* History of orthopedic or neurologic disorders to their intact limb, history of cardiovascular disease that prevents them from safely completing requested activities, unable to walk for 30 minutes at a time

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-07; Primary Completion 2019-08 (Actual); Study Completion 2019-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deanna H Gates, Ph.D., Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim J, Wensman J, Colabianchi N, Gates DH. The influence of powered prostheses on user perspectives, metabolics, and activity: a randomized crossover trial. J Neuroeng Rehabil. 2021 Mar 16;18(1):49. doi: 10.1186/s12984-021-00842-2. PMID 33726802

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began after initial approval from the University of Michigan IRB (July 2016). Participants were recruited through the University of Michigan Orthotics and Prosthetics Clinic by a study physician and study prosthetist in-person, through phone or email, or with flyers.
Pre-assignment Details: Participants were asked to complete both arms of the study. Before starting, participants were randomly enrolled in the dynamic response foot (unpowered prosthesis) or powered condition to start with. Some participants completed both arms while others only finished one of the arms.
Groups:
- Powered Ankle Prosthesis, Then Unpowered Prosthesis: In this condition, the participant was fitted with a powered prosthetic ankle by a certified prosthetist to start the study. The ankle is the BiOM which is manufactured by Bionx (which used to be named iWalk). This device was given 510(K) Exempt status by the FDA under (regulation number: 890.3500). Participants had at least one week to acclimate to the prosthesis. They then will wore the device for 2 weeks at home, while their activity was monitored. They then came to the lab for testing. The powered prosthesis was removed and their prescribed prosthetic foot was reattached to their existing socket. They then wore their prescribed prosthesis for 2 weeks, while their activity was monitored, before returning to the lab for testing.
- Unpowered Prosthesis, Then Powered Ankle Prosthesis: In this arm, participants will start in their clinically prescribed dynamic response foot. They first wore their prescribed prosthesis for 2 weeks, while their activity was monitored. They then came to the laboratory for testing. Participants were then fitted with a powered prosthetic ankle by a certified prosthetist. The ankle is the BiOM which is manufactured by Bionx (which used to be named iWalk). This device was given 510(K) Exempt status by the FDA under (regulation number: 890.3500). Participants had at least one week to acclimate to the prosthesis. They then will wore the device for 2 weeks at home, while their activity was monitored. They then came to the lab for testing. The powered prosthesis was removed and their prescribed prosthetic foot was reattached to their existing socket.
Period: First Intervention (3 Weeks)
Arm/Group | Powered Ankle Prosthesis, Then Unpowered Prosthesis | Unpowered Prosthesis, Then Powered Ankle Prosthesis
Started | 5 | 7
Received Intervention | 5 | 7
Completed | 4 | 6
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1
Period: Second Intervention (3 Weeks)
Arm/Group | Powered Ankle Prosthesis, Then Unpowered Prosthesis | Unpowered Prosthesis, Then Powered Ankle Prosthesis
Started | 4 | 6
Received Intervention | 4 | 6
Completed | 4 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: This group represents all participants enrolled in the study.
Arm/Group | All Study Participants
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.27 (13.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Metabolic Cost of Walking
Description: Metabolic costs will be measured using a portable metabolic system when participants walk on a treadmill at a fixed speed.
Time Frame: Testing took place after wearing the prostheses for two weeks
Population: Each participant wore both study prostheses. One participant was excluded from analysis as he was not able to reach steady-state energetics on a treadmill
Measure: Mean (Standard Deviation); unit: J/Nm
Groups:
- Unpowered Prosthesis: This condition is any unpowered prosthesis that was clinically prescribed to the patient
- BiOM Powered Prosthesis: This device is a prosthetic ankle which is battery powered and supplies active ankle power.
Arm/Group | Unpowered Prosthesis | BiOM Powered Prosthesis
Number analyzed (Participants) | 9 | 9
J/Nm | 0.409 (0.040) | 0.397 (0.078)
Statistical Analysis 1: Comparison: Unpowered Prosthesis vs BiOM Powered Prosthesis; The null hypothesis was that there would be no difference in metabolic costs between the two groups; Test type: Superiority; p = 0.585, t-test, 2 sided — Statistical significance was set a-priori at p<0.05

2. Primary Outcome: Total Steps Outside the Home Over a Two Week Period
Description: Activity data we be collected using activity monitors and GPS with both the regular prosthesis and the powered ankle prosthesis. Each activity monitoring period will last 2 weeks and will be done within in a 2 month period. Daily step count taken outside of the home, determined using an activity monitor and GPS device
Time Frame: 2 weeks
Population: Each participant in the study wore both prostheses
Measure: Mean (Standard Deviation); unit: steps
Groups:
- BiOM Powered Prostheis: This device is a prosthetic ankle which is battery powered and supplies active ankle power.
Arm/Group | Unpowered Prosthesis | BiOM Powered Prostheis
Number analyzed (Participants) | 10 | 10
steps | 2030 (1440) | 1640 (1100)
Statistical Analysis 1: Comparison: Unpowered Prosthesis vs BiOM Powered Prostheis; The null hypothesis was that there were no differences in the number of steps taken outside of the home for the two prostheses; Test type: Superiority; p = 0.452, t-test, 2 sided — Statistical significance was set a-priori at p<0.05

3. Primary Outcome: Quality of Life (QoL) on a Short-Form 36
Description: Participants completed the Medical Outcomes Study 36 Items Short-Form Health Survey (SF-36) after each condition. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability.
Time Frame: Questionnaire completed 2 weeks after wearing each prosthesis
Population: Each participant in the study wore both prostheses
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Unpowered Prosthesis | BiOM Powered Prosthesis
Number analyzed (Participants) | 10 | 10
scores on a scale
  Physical Component Score | 62.9 (17.5) | 59.4 (22)
  Mental Component Score | 63.6 (19.1) | 67.4 (24.0)
Statistical Analysis 1: Comparison: Unpowered Prosthesis vs BiOM Powered Prosthesis; Test type: Other — paired t-test of Physical component scores between the two conditions; p = 0.480, t-test, 2 sided — a prior threshold for significance was 0.05
Statistical Analysis 2: Comparison: Unpowered Prosthesis vs BiOM Powered Prosthesis; Mental Component Score; Test type: Superiority; p = 0.408, t-test, 2 sided — Statistical significance was set a-priori at p<0.05

4. Secondary Outcome: Prosthetic Evaluation Questionnaire (PEQ)
Description: Participants completed a survey to evaluate their prosthetic satisfaction (Prosthetic Evaluation Questionnaire) after each condition. Most questions in the PEQ use a visual analog scale format. Each visual analog scale is scored as a continuous numerical variable measured as the distance in millimeters from the left endpoint of the line (0 mm) to the point at which the respondent's mark crosses the line (up to 100 mm). The questions are all worded so that a higher number (toward the right) will correspond with a more positive response.
  Ambulation - Greater number = increased perceived ambulation Appearance - Greater number = better appearance Frustration - Greater number = less frustration Perceived Response - Greater number = increased perceived response Residual Limb Health - Greater number = better residual limb health Social burden - Greater number = less social burden Sounds - Greater number = less sound Utility - Greater
Time Frame: Questionnaire completed 2 weeks after wearing each prosthesis
Population: Each participant wore both study prostheses.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Unpowered Prosthesis | BiOM Powered Prosthesis
Number analyzed (Participants) | 10 | 10
scores on a scale
  Ambulation | 75.2 (18.3) | 84.0 (15.8)
  Appearance | 85.6 (9.58) | 80.6 (12.8)
  Frustration | 66.8 (29.7) | 84.8 (27.8)
  Perceived Response | 87.6 (20.7) | 97.1 (4.33)
  Residual Limb Health | 73.6 (19.4) | 79.9 (14.3)
  Social Burden | 85.2 (19.5) | 91.6 (15.3)
  Sounds | 71.4 (27.1) | 57.2 (31.5)
  Utility | 73.1 (14.8) | 74.4 (16.7)
  Well-Being | 72.9 (26.9) | 79.2 (22.0)
Statistical Analysis 1: Comparison: Unpowered Prosthesis vs BiOM Powered Prosthesis; Ambulation Score; Test type: Superiority; p = 0.058, t-test, 2 sided — Statistical significance was set a-priori at p<0.05
Statistical Analysis 2: Comparison: Unpowered Prosthesis vs BiOM Powered Prosthesis; Appearance Score; Test type: Other — paired t-test between conditions; p = .123, t-test, 2 sided — Statistical significance was set a-priori at p<0.05
Statistical Analysis 3: Comparison: Unpowered Prosthesis vs BiOM Powered Prosthesis; Frustration Score; Test type: Other — paired t-test between conditions; p = .052, t-test, 2 sided — Statistical significance was set a-priori at p<0.05
Statistical Analysis 4: Comparison: Unpowered Prosthesis vs BiOM Powered Prosthesis; Perceived Response Score; Test type: Other — paired t-test between conditions; p = .188, t-test, 2 sided — Statistical significance was set a-priori at p<0.05
Statistical Analysis 5: Comparison: Unpowered Prosthesis vs BiOM Powered Prosthesis; Residual Limb Health Score; Test type: Other — paired t-test between conditions; p = .336, t-test, 2 sided — Statistical significance was set a-priori at p<0.05
Statistical Analysis 6: Comparison: Unpowered Prosthesis vs BiOM Powered Prosthesis; Social Burden Score; Test type: Other — paired t-test between conditions; p = .043, t-test, 2 sided — Statistical significance was set a-priori at p<0.05
Statistical Analysis 7: Comparison: Unpowered Prosthesis vs BiOM Powered Prosthesis; Sounds Score; Test type: Other — paired t-test between conditions; p = .391, t-test, 2 sided — Statistical significance was set a-priori at p<0.05
Statistical Analysis 8: Comparison: Unpowered Prosthesis vs BiOM Powered Prosthesis; Utility Score; Test type: Superiority — paired t-test between conditions; p = .799, t-test, 2 sided — Statistical significance was set a-priori at p<0.05
Statistical Analysis 9: Comparison: Unpowered Prosthesis vs BiOM Powered Prosthesis; Well-Being; Test type: Superiority; p = .173, t-test, 2 sided — Statistical significance was set a-priori at p<0.05

5. Secondary Outcome: Muscle Activity in the Lower Limb
Description: Participants walk on a treadmill while muscle activity from various lower limb muscles are monitored using electromyography. We calculated the integrated EMG (iEMG) for each muscle collected as the total activity in that muscle as a percentage of the maximum signal.
Time Frame: Testing took place after the participant wore the prosthesis for 2 weeks
Population: Each participant wore both study prostheses
Measure: Mean (Standard Deviation); unit: percentage of maximum signal
Arm/Group | Unpowered Prosthesis | BiOM Powered Prosthesis
Number analyzed (Participants) | 9 | 9
percentage of maximum signal
  Intact side biceps femoris | 24.3 (5.07) | 24.1 (8.83)
  Intact side rectus femoris | 25.3 (4.06) | 28.7 (14.1)
  Intact side soleus | 29.9 (6.47) | 28.6 (9.11)
  Intact side tibialis anterior | 28.4 (10.2) | 30.4 (7.99)
  Residual side biceps femoris | 27.8 (10.8) | 25.9 (8.70)
  Residual side rectus femoris | 38.3 (12.2) | 41.3 (9.01)
Statistical Analysis 1: Comparison: Unpowered Prosthesis vs BiOM Powered Prosthesis; Intact Side Biceps Femoris; Test type: Other — paired t-test between conditions; p = 0.655, t-test, 2 sided — Statistical significance was set a-priori at p<0.05
Statistical Analysis 2: Comparison: Unpowered Prosthesis vs BiOM Powered Prosthesis; Intact Side Rectus Femoris; Test type: Other — paired t-test between conditions; p = .281, t-test, 2 sided — Statistical significance was set a-priori at p<0.05
Statistical Analysis 3: Comparison: Unpowered Prosthesis vs BiOM Powered Prosthesis; Intact Side Soleus; Test type: Other — paired t-test between conditions; p = .844, t-test, 2 sided — Statistical significance was set a-priori at p<0.05
Statistical Analysis 4: Comparison: Unpowered Prosthesis vs BiOM Powered Prosthesis; Intact Side Tibialis Anterior; Test type: Other — paired t-test between conditions; p = .110, t-test, 2 sided — Statistical significance was set a-priori at p<0.05
Statistical Analysis 5: Comparison: Unpowered Prosthesis vs BiOM Powered Prosthesis; Residual Side Biceps Femoris; Test type: Other — paired t-test between conditions; p = .394, t-test, 2 sided — Statistical significance was set a-priori at p<0.05
Statistical Analysis 6: Comparison: Unpowered Prosthesis vs BiOM Powered Prosthesis; Residual Side Rectus Femoris; Test type: Superiority; p = .141, t-test, 2 sided — Statistical significance was set a-priori at p<0.05

6. Secondary Outcome: Time to Fatigue
Description: Participants walk on a treadmill at a fast speed until they felt they can no longer continue. The time to fatigue was recorded.
Time Frame: Testing took place after wearing the prostheses for two weeks
Population: Each participant wore both study prostheses
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Unpowered Prosthesis | BiOM Powered Prosthesis
Number analyzed (Participants) | 10 | 10
minutes | 14.7 (12.1) | 13.2 (10.8)
Statistical Analysis 1: Comparison: Unpowered Prosthesis vs BiOM Powered Prosthesis; Test type: Superiority; p = 0.212, t-test, 2 sided — Statistical significance was set a-priori at p<0.05

ADVERSE EVENTS:
Time Frame: Adverse events were monitored through study completion for each participant, which was approximately 3 months time.
Description: If an adverse event were to occur, it would be reported to the University of Michigan IRB and study sponsor for review.
Groups:
- Powered Ankle Prosthesis: In this condition, the participant is fitted with a powered prosthetic ankle by a certified prosthetist. The ankle is the BiOM which is manufactured by Bionx (which used to be named iWalk). This device was given 510(K) Exempt status by the FDA under (regulation number: 890.3500). After accommodation, participants wore the device for 2 weeks.
  Powered ankle prosthesis: This device is a commercially available powered ankle prosthesis, (BioM, Bionx, Bedford, MA) which was given FDA device exempt status.
  We monitored for adverse events the entire time the participant had the device at home for accommodation and monitoring (~ 3 weeks)
- Unpowered Prosthesis: In this arm, participants will wear their clinically prescribed dynamic response foot (unpowered prosthesis). This period is 2 weeks long.
  Dynamic Response Foot: This condition is a sham condition as the participant will wear the prosthesis they were clinically prescribed and usually wear.
  We monitored for adverse events the entire time the person wore their device at home and were monitored (2 weeks).
Arm/Group | Powered Ankle Prosthesis | Unpowered Prosthesis
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-02): https://cdn.clinicaltrials.gov/large-docs/82/NCT02828982/Prot_SAP_000.pdf